CLINICAL TRIAL: NCT01028417
Title: A Randomized Controlled Trial To Determine If Thoracoscopic Resection Of Subcentimetre Lung Nodules After Localization Using Percutaneously Inserted Platinum Microcoils Under CT Guidance Reduces Rate Of Conversion To Open Thoracotomy From 50% To 10%
Brief Title: Study to See if Microcoil Insertion Reduces the Rate of Open Thoracotomy for Removal of Lung Nodules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H09-02265
Record Dates: First submitted 2009-12-03; First posted 2009-12-09 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: subcentimetre nodules
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1 receives the intervention - insertion of platinum microcoil followed by nodule excision
  Interventions: Device: Platinum microcoil
- Group 2 (No Intervention): Group 2 receives the standard of care - nodule excision, but without the microcoil insertion

INTERVENTIONS:
Device: Platinum microcoil — Coil Name: Vortx-18, Diamond Shape, Boston Scientific, Cork, Ireland; Coil Description: 80 mm long, fibre coated 0.018 inch diameter platinum microcoil
  Arms: Group 1

SUMMARY:
LAY ABSTRACT

1. Statement of the health problem or issue: Of the estimated 24,000 Canadians who will be diagnosed with lung cancer in 2008, 21,000 will die of their disease. Based on this cancer incidence and survival data, the most promising current strategy for improving outcome is screening and early detection. It is suggested that if lesions are discovered at an earlier stage of disease, they will have a higher likelihood of being treatable and therefore, survival will be improved. CT detection of growing small lung nodules, many of which are non-cancerous (benign), raises the possibility of lung cancer and thus causes anxiety in patients and referring clinicians. Unfortunately, confident separation of benign from malignant small lung nodules cannot be reliably achieved using CT or PET criteria. Pathologic diagnosis using needle or excision biopsy is usually required.

   Excision biopsy removes the entire nodule at one setting and eliminates the sampling error associated with needle biopsy, making it appealing to physicians and patients. To reduce post-operative pain and breathing difficulties, excision biopsy is often performed using minimally invasive surgery (video assisted thoracoscopic surgery, VATS). Finding small pulmonary nodules is often difficult with the minimally invasive camera (VATS) and a bigger incision (thoracotomy) is necessary in more than 60% of our patients.

   We recently developed a technique of using platinum micro-coils, which are inserted in the lung nodule using CT guidance, to locate the nodule with fluoroscopy and then excise it with VATS. We have completed a pilot study (n=75 nodules; 69 patients) to determine the effectiveness of this technique. Seventy three (97%) 4-24-mm nodules were successfully removed at fluoroscopically guided VATS excision.
2. Objective of your project: To improve our ability to successfully excise small growing lung nodules with minimally invasive VATS surgery using CT guided micro-coil localization techniques.
3. How will you undertake your work? We propose to conduct a randomized controlled trial to determine if the use of CT guided platinum microcoil markers for VATS excision of subcentimetre pulmonary nodules can reduce the rate of conversion to open thoracotomy from 50% to 10%.
4. What is unique/innovative about your project? New image guided minimally invasive surgical technique for removing early growing cancers was developed at the Vancouver General Hospital and the University of British Columbia. This has been published in peer-reviewed journals and can potentially allow us to accurately locate and excise suspicious lung nodules
5. Relevance to Lung Association's mission statement? Lung cancer remains a major health problem in Canada. Early detection and screening programs allow for discovery of nodules when they are still very small and therefore, likely curable. Excision biopsy removes the entire nodule at one setting and eliminates the sampling error associated with needle biopsy, making it appealing to patients and physicians. To reduce post operative morbidity, costs and volume of lung removed, excision biopsy is often performed using video assisted thoracoscopic surgery (VATS) techniques. Using a pilot project grant from the BC Lung Association we have developed a new technique that allows preoperative CT marking of the nodule and minimally invasive removal of the lesion. We hope that this technique will allow earlier treatment of lung cancers and improve survival in this devastating disease.

DETAILED DESCRIPTION:
Intervention Description:

The pre-operative CT scan will be reviewed by the surgeon with the radiologist to determine if the nodule can be excised using thoracoscopic staple wedge techniques. After informed consent, the patient will be seen by an anesthesiologist to determine risks and benefits of a general anesthetic. The patient will initially come to the CT scanner suite in the radiology department. The CT guided percutaneous microcoil nodule localization procedure, will be performed consciously under local anaesthesia Using sterile technique and local anesthetic, a biopsy needle (22 gauge) pre-loaded with an 6 cm long platinum microcoil will be placed 10mm deep to the suspicious pulmonary nodule using CT guidance. The coil will be deployed such that one end will be adjacent to the nodule and the other end will lie free on the: lung surface. The patient will be transferred to the Laurel OR where they will be placed under general anesthesia with a double lumen endotracheal tube in order to allow collapse of the involved lung during the thoracoscopic excision of the marked lung nodule. The patient's blood pressures, oxygen levels, pulse and ECG will be monitored. The thoracoscopic excision of the nodule will be performed using the microcoil as a localizing device. Using the preoperative CT scan, the study surgeon will mark the insertion sites for thoracoscopic instruments. Instruments for video-assisted thoracoscopy include a rigid 5 mm thoracoscope, a light source, a video-camera and monitor, and 5 mm grasping forceps. The patient will be draped. A 5mm thoracoscopic port is inserted into the thorax percutaneously and the lung is examined with the thoracoscope. The nodule location will be identified by the end of the microcoil that sits on the surface of the lung. A second 5 mm port is put in place and the end of the microcoil grasped under thoracoscopic visualization. Multiple endoscopic are placed via a third 12mm port and the nodule and coil are completely excised under fluoroscopic guidance. The resected nodule is placed in an endoscopic bag and brought out through the large port site. If the lesion cannot be excised by the VATS technique the patient will undergo an open rib spreading thoracotomy for excision of the marked nodule. The indications for thoracotomy at this time are:poor visualization of the lung, pleural symphysis with scarring, uncontrollable bleeding or inability to completely resect the lesion with the thoracoscopic endostapler.

The specimen is sent for frozen section pathological examination. If the lesion is benign the thoracic cavity is irrigated with saline and a small chest tube is put in place and attached to under water drainage. The incisions are then closed and the lung is re-expanded. The patient is then transported to the post-anesthetic room similar to other patients undergoing general anesthesia. If the lesion is a non-small cell cancer of the lung the patient may undergo a sampling of lymph nodes at that time followed by formal lobectomy. If the patient has inadequate pulmonary function to tolerate a lobectomy and the lesion has been completely excised the surgeon may choose to stop the operation at that time and follow the patient.

ELIGIBILITY:
Inclusion Criteria: Patients will be evaluated for eligibility using the following criteria:

* All newly diagnosed patients with small lung nodules < 1cm that require excision with no history of prior ipsilateral thoracotomy.
* The nodules must be located in parts of the lung that are amenable to thoracoscopic wedge excision of the nodules.The external surface of the lesion must be at least 2 cm from the major pulmonary arteries, veins, and main bronchi to allow safe and adequate thoracoscopic excision of the lesion.
* Patients must be mentally competent to give written, informed consent
* Patients must be capable of independently completing standard English-language QOL instruments.

Exclusion Criteria:

* Patients will be excluded from the trial if they do not consent to participate in the study, or if the radiologist and surgeon agree that the nodule is located too centrally to be safely excised using thoracoscopic wedge techniques.
* Patients with more than three nodules will be excluded from the study.
* Patients with a positive diagnosis of non-small cell lung cancer obtained from sputum cytology, bronchoscopy, or CT guided needle biopsy will be excluded from the study.
* If the patient is excluded, he/she will receive the current standard treatment, which may include needle biopsy, continued observation of the nodule at three to six monthly intervals, or excisional surgery (thoracoscopy or open thoracotomy).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
conversion to open thoracotomy | final surgery June15, 2012

SECONDARY OUTCOMES:
the quality of life using well-validated quality of life instruments | last date July 15, 2013
the preoperative, intraoperative and postoperative costs | end: July 15, 2013
the perioperative morbidity and mortality | last date June 15, 2012

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finley, MD, Principal Investigator — University of British Columbia; John Mayo, Study Director — University of British Columbia; Joanne Clifton, Study Director — University of British Columbia; John Yee, Study Director — University of British Columbia; Ken Evans, Study Director — University of British Columbia; John English, Study Director — University of British Columbia; Larry Lynd, Study Director — University of British Columbia
Locations (1):
- Vancouver General Hospital - Diamond Pavilion, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Finley RJ, Mayo JR, Grant K, Clifton JC, English J, Leo J, Lam S. Preoperative computed tomography-guided microcoil localization of small peripheral pulmonary nodules: a prospective randomized controlled trial. J Thorac Cardiovasc Surg. 2015 Jan;149(1):26-31. doi: 10.1016/j.jtcvs.2014.08.055. Epub 2014 Sep 16. PMID 25293355